CLINICAL TRIAL: NCT00293930
Title: A Study to Assess the Safety and Effectiveness of Tacrolimus Cream in the Treatment of Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-0-205
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2007-12-24 (Estimated); Status verified 2007-12

CONDITIONS: Psoriasis
Keywords: Treatment Outcome; Tacrolimus; Safety; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
A study to assess the safety and effectiveness of tacrolimus cream in the treatment of psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of plaque psoriasis

Exclusion Criteria:

* Skin disorder other than plaque psoriasis in the areas to be treated.
* Disease on only elbows, knees, and scalp

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Rico, MD, Study Director — Astellas Pharma US, Inc.
Locations (32):
- United States (26):
  - Hot Springs, Arkansas
  - San Diego, California
  - San Francisco, California
  - Longmont, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Newnan, Georgia
  - Evansville, Indiana
  - South Bend, Indiana
  - Iowa City, Iowa
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Bryan, Texas
  - Dallas, Texas
  - Galveston, Texas
  - Burlington, Vermont
  - Lynchburg, Virginia
  - Dayton, Washington
  - Madison, Wisconsin
- Canada (6):
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - North Bay, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Saskatoon, Saskatchewan